CLINICAL TRIAL: NCT00843115
Title: Ecological Perspective On The Efficacy And Tolerability Of Donepezil In A Routine Clinical Practice: A Patient Centered Observational Study
Brief Title: Observational Study Of Donepezil In Routine Clinical Practice
Status: Terminated | Type: Observational
Why Stopped: See Detailed Description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: NRA2500065; ECO STUDY
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Results first posted 2009-06-02 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-02

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease, naturalistic study
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational: This study was non-interventional and simply followed for 3 months patients initiating a treatment with donepezil
  Interventions: Other: donepezil

INTERVENTIONS:
Other: donepezil — Routine clinical practice of prescribing donepezil as per the Canadian label. No drug was supplied as part of this study
  Other Names: Aricept

SUMMARY:
To characterize the comorbidities and medications of patients treated with donepezil in a routine clinical practice and to verify the therapeutic response of these patients.

DETAILED DESCRIPTION:
This trial was terminated prematurely on December 31, 2007 due to difficulties in enrolling patients in the study. There were no safety or efficacy concerns regarding the study in the decision to terminate the trial.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV criteria for the clinical diagnosis of mild to moderate Alzheimer's Disease with or without other etiologies of dementia
* Mini Mental Status Examination score of 10-26

Exclusion Criteria:

* Contraindication as stated in the Canadian label for donepezil
* Subjects treated with medication for dementia within 30 days prior to baseline

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Alzheimer's Disease with or without other etiologies of dementia
Sampling Method: Non-Probability Sample
Enrollment: 370 (Actual)
Dates: Start 2007-02; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=NRA2500065&StudyName=Observational%20Study%20Of%20Donepezil%20In%20Routine%20Clinical%20Practice

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a non interventional study conducted at 62 sites in Canada.
Pre-assignment Details: Subjects had a diagnosis of mild to moderate Alzheimer's Disease with or without other etiologies of dementia.
Groups:
- Donepezil: As per physician prescription
Period: Overall Study
Arm/Group | Donepezil
Started | 370
Completed | 304
Not Completed | 66
Not completed — Death | 4
Not completed — Adverse Event | 30
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 17
Not completed — Family wanted meds stopped | 1
Not completed — Family does not want continuation | 1
Not completed — Patient forgot to take meds | 1
Not completed — Does not meet entrance criteria | 1
Not completed — Physician Decision | 1
Not completed — Family discontinued meds | 1
Not completed — patient took for 2 days then stopped | 1
Not completed — patient never took the medication | 1
Not completed — hospitalized due to deterioration | 1
Not completed — week 12 not done | 1
Not completed — Syndrome De Glissement | 1

BASELINE CHARACTERISTICS:
Arm/Group | Donepezil
Number analyzed (Participants) | 370
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.1 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172
  Male | 198

OUTCOME MEASURES:

1. Primary Outcome: All Subjects Improved/Stabilized or Worsened for Cognitive Activation in Top Symptom Checklist (TOPS) Alzheimer's Disease Assessment
Description: Cognitive Activation symptom in TOPS checklist: Number of subjects Improved/Stabilized or Worsened. TOPS Ratings compared at baseline & Week 12. No symptoms=1, Emergence of symptoms=2, Symptoms Increased=3, Stable=4, Symptoms decreased=5, Cessation of Symptoms=6. Ratings recoded to Categories: Improved/Stabilized=4,5,6; Worsened=2,3.
Time Frame: Baseline and Week 12
Population: Intent to Treat (ITT): All Subjects who did not have a response for post baseline assessment were not included in analysis.
Measure: Number; unit: participants
Arm/Group | Donepezil
Number analyzed (Participants) | 322
participants
  Improved or Stabilized | 196
  Worsened | 36
  Missing/Not Applicable | 90
Statistical Analysis 1: Comparison: Donepezil; null hypothesis: the proportion of subjects who improved or stabilized, among those who had the symptom at baseline, is less than or equal to 0.5; the alternative hypothesis: this proportion is greater than 0.5; Test type: Superiority or Other; p < 0.0001, Binomial test of proportions; Holms multiplicity adjustment (Stepdown Bonferroni) for statistical significance of each p-value, while controlling experiment wise error rate at 0.05

2. Primary Outcome: All Subjects Improved/Stabilized or Worsened for Attention in Top Symptom Checklist (TOPS) Alzheimer's Disease Assessment
Description: Attention symptom in TOPS checklist: Number of subjects Improved/Stabilized or Worsened. TOPS Ratings compared at baseline and Week 12. No symptoms=1, Emergence of symptoms=2, Symptoms Increased=3, Stable=4, Symptoms decreased=5, Cessation of Symptoms=6. Ratings recoded to Improved/Stabilized=4,5,6; Worsened=2,3.
Time Frame: Baseline and Week 12
Population: Intent to Treat (ITT) : All subjects who did not have a response for post baseline assessment were not included in analysis.
Measure: Number; unit: Participants
Arm/Group | Donepezil
Number analyzed (Participants) | 322
Participants
  Improved or Stabilized | 202
  Worsened | 31
  Missing/Not Applicable | 89
Statistical Analysis 1: Comparison: Donepezil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Binomial test of proportions; Holms multiplicity adjustment Stepdown Bonferroni) for statistical significance of each p-value, while controlling experiment wise error rate at 0.05

3. Primary Outcome: All Subjects Improved/Stabilized or Worsened for Repetitiveness in Top Symptom Checklist (TOPS) Alzheimer's Disease Assessment
Description: Repetitiveness symptom in TOPS checklist: Number of subjects Improved/Stabilized or Worsened. TOPS Ratings compared at baseline & Week 12. No symptoms=1, Emergence of symptoms=2, Symptoms Increased=3, Stable=4, Symptoms decreased=5, Cessation of Symptoms=6. Ratings recoded to Categories: Improved/Stabilized=4,5,6; Worsened=2,3.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Donepezil
Number analyzed (Participants) | 322
Participants
  Improved or Stabilized | 195
  Worsened | 32
  Missing/Not Applicable | 95
Statistical Analysis 1: Comparison: Donepezil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Binomial test of proportions; [statistical method as in outcome 1, analysis 1]

4. Primary Outcome: All Subjects Improved/Stabilized or Worsened for Remembering in Top Symptom Checklist (TOPS) Alzheimer's Disease Assessment
Description: Remembering symptom in TOPS checklist: Number of subjects Improved/Stabilized or Worsened. TOPS Ratings compared at baseline & Week 12. No symptoms=1, Emergence of symptoms=2, Symptoms Increased=3, Stable=4, Symptoms decreased=5, Cessation of Symptoms=6. Ratings recoded toCategories: Improved/Stabilized=4,5,6; Worsened=2,3.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Donepezil
Number analyzed (Participants) | 322
participants
  Improved or Stabilized | 231
  Worsened | 44
  Missing/Not Applicable | 47
Statistical Analysis 1: Comparison: Donepezil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Binomial test of proportions; [statistical method as in outcome 1, analysis 1]

5. Primary Outcome: All Subjects Improved/Stabilized or Worsened for Temporal Orientation in Top Symptom Checklist (TOPS) Alzheimer's Disease Assessment
Description: Temporal Orientation symptom in TOPS checklist: Number of subjects Improved/Stabilized or Worsened. TOPS Ratings compared at baseline & Week 12. No symptoms=1, Emergence of symptoms=2, Symptoms Increased=3, Stable=4, Symptoms decreased=5, Cessation of Symptoms=6. Ratings recoded to Categories: Improved/Stabilized=4,5,6; Worsened=2,3.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Donepezil
Number analyzed (Participants) | 322
Participants
  Improved or Stabilized | 209
  Worsened | 39
  Missing/Not Applicable | 74
Statistical Analysis 1: Comparison: Donepezil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Binomial test of proportions; [statistical method as in outcome 1, analysis 1]

6. Primary Outcome: All Subjects Improved/Stabilized or Worsened for Asphasia in Top Symptom Checklist (TOPS) Alzheimer's Disease Assessment
Description: Asphasia symptom in TOPS checklist: Number of subjects Improved/Stabilized or Worsened. TOPS Ratings compared at baseline & Week 12. No symptoms=1, Emergence of symptoms=2, Symptoms Increased=3, Stable=4, Symptoms decreased=5, Cessation of Symptoms=6. Ratings recoded toCategories: Improved/Stabilized=4,5,6; Worsened=2,3.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Donepezil
Number analyzed (Participants) | 322
participants
  Improved or Stabilized | 190
  Worsened | 28
  Missing/Not Applicable | 104
Statistical Analysis 1: Comparison: Donepezil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Binomial test of proportions; [statistical method as in outcome 1, analysis 1]

7. Primary Outcome: All Subjects Improved/Stabilized or Worsened for Spatial Orientation in Top Symptom Checklist (TOPS) Alzheimer's Disease Assessment
Description: Spatial Orientation symptom in TOPS checklist: Number of subjects Improved/Stabilized or Worsened. TOPS Ratings compared at baseline & Week 12. No symptoms=1, Emergence of symptoms=2, Symptoms Increased=3, Stable=4, Symptoms decreased=5, Cessation of Symptoms=6. Ratings recoded to categories: Improved/Stabilized=4,5,6; Worsened=2,3
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Donepezil
Number analyzed (Participants) | 322
participants
  Improved or Stabilized | 201
  Worsened | 25
  Missing/Not Applicable | 96
Statistical Analysis 1: Comparison: Donepezil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Binomial test of proportions; [statistical method as in outcome 1, analysis 1]

8. Primary Outcome: All Subjects Improved/Stabilized or Worsened for Judgment in Top Symptom Checklist (TOPS) Alzheimer's Disease Assessment
Description: Judgment symptom in TOPS checklist: Number of subjects Improved/Stabilized or Worsened. TOPS Ratings compared at baseline & Week 12. No symptoms=1, Emergence of symptoms=2, Symptoms Increased=3, Stable=4, Symptoms decreased=5, Cessation of Symptoms=6. Ratings recoded to Categories: Improved/Stabilized=4,5,6; Worsened=2,3.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Donepezil
Number analyzed (Participants) | 322
participants
  Improved or Stabilized | 206
  Worsened | 30
  Missing/Not Applicable | 86
Statistical Analysis 1: Comparison: Donepezil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Binomial test of proportions; [statistical method as in outcome 1, analysis 1]

9. Primary Outcome: All Subjects Improved/Stabilized or Worsened for Insight in Top Symptom Checklist (TOPS) Alzheimer's Disease Assessment
Description: Insight symptom in TOPS checklist: Number of subjects Improved/Stabilized or Worsened. TOPS Ratings compared at baseline & Week 12. No symptoms=1, Emergence of symptoms=2, Symptoms Increased=3, Stable=4, Symptoms decreased=5, Cessation of Symptoms=6. Ratings recoded to Categories: Improved/Stabilized=4,5,6; Worsened=2,3.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Donepezil
Number analyzed (Participants) | 322
participants
  Improved or Stabilized | 209
  Worsened | 34
  Missing/Not Applicable | 79
Statistical Analysis 1: Comparison: Donepezil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Binomial test of proportions; [statistical method as in outcome 1, analysis 1]

10. Primary Outcome: All Subjects Improved/Stabilized or Worsened for Leisure in Top Symptom Checklist (TOPS) Alzheimer's Disease Assessment
Description: Leisure symptom in TOPS checklist: Number of subjects Improved/Stabilized or Worsened. TOPS Ratings compared at baseline & Week 12. No symptoms=1, Emergence of symptoms=2, Symptoms Increased=3, Stable=4, Symptoms decreased=5, Cessation of Symptoms=6. Ratings recoded to Categories: Improved/Stabilized=4,5,6; Worsened=2,3.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Donepezil
Number analyzed (Participants) | 322
participants
  Improved or Stabilized | 205
  Worsened | 28
  Missing/Not Applicable | 89
Statistical Analysis 1: Comparison: Donepezil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Binomial test of proportions; [statistical method as in outcome 1, analysis 1]

11. Primary Outcome: All Subjects Improved/Stabilized or Worsened for Domestic Activities in Top Symptom Checklist (TOPS) Alzheimer's Disease Assessment
Description: Domestic Activities symptom in TOPS checklist: Number of subjects Improved/Stabilized or Worsened. TOPS Ratings compared at baseline & Week 12. No symptoms=1, Emergence of symptoms=2, Symptoms Increased=3, Stable=4, Symptoms decreased=5, Cessation of Symptoms=6. Ratings recoded to Categories: Improved/Stabilized=4,5,6; Worsened=2,3.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Donepezil
Number analyzed (Participants) | 322
participants
  Improved or Stabilized | 198
  Worsened | 23
  Missing/Not Applicable | 101
Statistical Analysis 1: Comparison: Donepezil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Binomial test of proportions; [statistical method as in outcome 1, analysis 1]

12. Primary Outcome: All Subjects Improved/Stabilized or Worsened for Hygiene in Top Symptom Checklist (TOPS) Alzheimer's Disease Assessment
Description: Hygiene symptom in TOPS checklist: Number of subjects Improved/Stabilized or Worsened. TOPS Ratings compared at baseline & Week 12. No symptoms=1, Emergence of symptoms=2, Symptoms Increased=3, Stable=4, Symptoms decreased=5, Cessation of Symptoms=6. Ratings recoded to Categories: Improved/Stabilized=4,5,6; Worsened=2,3.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Donepezil
Number analyzed (Participants) | 322
participants
  Improved or Stabilized | 168
  Worsened | 23
  Missing/Not Applicable | 131
Statistical Analysis 1: Comparison: Donepezil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Binomial test of proportions; [statistical method as in outcome 1, analysis 1]

13. Primary Outcome: All Subjects Improved/Stabilized or Worsened for Dressing in Top Symptom Checklist (TOPS) Alzheimer's Disease Assessment
Description: Dressing symptom in TOPS checklist: Number of subjects Improved/Stabilized or Worsened. TOPS Ratings compared at baseline & Week 12. No symptoms=1, Emergence of symptoms=2, Symptoms Increased=3, Stable=4, Symptoms decreased=5, Cessation of Symptoms=6. Ratings recoded to Categories: Improved/Stabilized=4,5,6; Worsened=2,3.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Donepezil
Number analyzed (Participants) | 322
participants
  Improved or Stabilized | 152
  Worsened | 23
  Missing/Not Applicable | 147
Statistical Analysis 1: Comparison: Donepezil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Binomial test of proportions; [statistical method as in outcome 1, analysis 1]

14. Primary Outcome: All Subjects Improved/Stabilized or Worsened for Telephoning in Top Symptom Checklist (TOPS) Alzheimer's Disease Assessment
Description: Telephoning symptom in TOPS checklist: Number of subjects Improved/Stabilized or Worsened. TOPS Ratings compared at baseline & Week 12. No symptoms=1, Emergence of symptoms=2, Symptoms Increased=3, Stable=4, Symptoms decreased=5, Cessation of Symptoms=6. Ratings recoded to Categories: Improved/Stabilized=4,5,6; Worsened=2,3.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Donepezil
Number analyzed (Participants) | 322
participants
  Improved or Stabilized | 190
  Worsened | 16
  Missing/Not Applicable | 116
Statistical Analysis 1: Comparison: Donepezil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Binomial test of proportions; [statistical method as in outcome 1, analysis 1]

15. Primary Outcome: All Subjects Improved/Stabilized or Worsened for Agitation in Top Symptom Checklist (TOPS) Alzheimer's Disease Assessment
Description: Agitation symptom in TOPS checklist: Number of subjects Improved/Stabilized or Worsened. TOPS Ratings compared at baseline & Week 12. No symptoms=1, Emergence of symptoms=2, Symptoms Increased=3, Stable=4, Symptoms decreased=5, Cessation of Symptoms=6. Ratings recoded to Categories: Improved/Stabilized=4,5,6; Worsened=2,3.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Donepezil
Number analyzed (Participants) | 322
participants
  Improved or Stabilized | 157
  Worsened | 23
  Missing/Not Applicable | 142
Statistical Analysis 1: Comparison: Donepezil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Binomial test of proportions; [statistical method as in outcome 1, analysis 1]

16. Primary Outcome: All Subjects Improved/Stabilized or Worsened for Mood in Top Symptom Checklist (TOPS) Alzheimer's Disease Assessment
Description: Mood symptom in TOPS checklist: Number of subjects Improved/Stabilized or Worsened. TOPS Ratings compared at baseline & Week 12. No symptoms=1, Emergence of symptoms=2, Symptoms Increased=3, Stable=4, Symptoms decreased=5, Cessation of Symptoms=6. Ratings recoded to Categories: Improved/Stabilized=4,5,6; Worsened=2,3.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Donepezil
Number analyzed (Participants) | 322
participants
  Improved or Stabilized | 187
  Worsened | 38
  Missing/Not Applicable | 97
Statistical Analysis 1: Comparison: Donepezil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Binomial test of proportions; [statistical method as in outcome 1, analysis 1]

17. Primary Outcome: All Subjects Improved/Stabilized or Worsened for Anxiety in Top Symptom Checklist (TOPS) Alzheimer's Disease Assessment
Description: Anxiety symptom in TOPS checklist: Number of subjects Improved/Stabilized or Worsened. TOPS Ratings compared at baseline & Week 12. No symptoms=1, Emergence of symptoms=2, Symptoms Increased=3, Stable=4, Symptoms decreased=5, Cessation of Symptoms=6. Ratings recoded to Categories: Improved/Stabilized=4,5,6; Worsened=2,3.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Donepezil
Number analyzed (Participants) | 322
participants
  Improved or Stabilized | 195
  Worsened | 37
  Missing/Not Applicable | 90
Statistical Analysis 1: Comparison: Donepezil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Binomial test of proportions; [statistical method as in outcome 1, analysis 1]

18. Primary Outcome: All Subjects Improved/Stabilized or Worsened for Delusions in Top Symptom Checklist (TOPS) Alzheimer's Disease Assessment
Description: Delusions symptom in TOPS checklist: Number of subjects Improved/Stabilized or Worsened. TOPS Ratings compared at baseline & Week 12. No symptoms=1, Emergence of symptoms=2, Symptoms Increased=3, Stable=4, Symptoms decreased=5, Cessation of Symptoms=6. Ratings recoded to Categories: Improved/Stabilized=4,5,6; Worsened=2,3.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Donepezil
Number analyzed (Participants) | 322
participants
  Improved or Stabilized | 139
  Worsened | 16
  Missing/Not Applicable | 167
Statistical Analysis 1: Comparison: Donepezil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Binomial test of proportions; [statistical method as in outcome 1, analysis 1]

19. Primary Outcome: All Subjects Improved/Stabilized or Worsened for Apathy in Top Symptom Checklist (TOPS) Alzheimer's Disease Assessment
Description: Apathy symptom in TOPS checklist: Number of subjects Improved/Stabilized or Worsened. TOPS Ratings compared at baseline & Week 12. No symptoms=1, Emergence of symptoms=2, Symptoms Increased=3, Stable=4, Symptoms decreased=5, Cessation of Symptoms=6. Ratings recoded to Categories: Improved/Stabilized=4,5,6; Worsened=2,3.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Donepezil
Number analyzed (Participants) | 322
participants
  Improved or Stabilized | 187
  Worsened | 27
  Missing/Not Applicable | 108
Statistical Analysis 1: Comparison: Donepezil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Binomial test of proportions; Holms multiplicity adjustment (Stepdown Bonferroni) for statistical significance of each p-value, while controlling experiment wise error rate @ 0.05

20. Primary Outcome: All Subjects Improved/Stabilized or Worsened for Caregiver in Top Symptom Checklist (TOPS) Alzheimer's Disease Assessment
Description: Caregiver symptom in TOPS checklist: Number of subjects Improved/Stabilized or Worsened. TOPS Ratings compared at baseline & Week 12. No symptoms=1, Emergence of symptoms=2, Symptoms Increased=3, Stable=4, Symptoms decreased=5, Cessation of Symptoms=6. Ratings recoded to Categories: Improved/Stabilized=4,5,6; Worsened=2,3.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Donepezil
Number analyzed (Participants) | 322
participants
  Improved or Stabilized | 213
  Worsened | 30
  Missing/Not Applicable | 79
Statistical Analysis 1: Comparison: Donepezil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Binomial test of proportions; [statistical method as in outcome 1, analysis 1]

21. Primary Outcome: All Subjects Improved/Stabilized or Worsened for Severity in Top Symptom Checklist (TOPS) Alzheimer's Disease Assessment
Description: Severity symptom in TOPS checklist: Number of subjects Improved/Stabilized or Worsened. TOPS Ratings compared at baseline & Week 12. No symptoms=1, Emergence of symptoms=2, Symptoms Increased=3, Stable=4, Symptoms decreased=5, Cessation of Symptoms=6. Ratings recoded to Categories: Improved/Stabilized=4,5,6; Worsened=2,3.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Donepezil
Number analyzed (Participants) | 322
participants
  Improved or Stabilized | 233
  Worsened | 40
  Missing/Not Applicable | 49
Statistical Analysis 1: Comparison: Donepezil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Binomial test of proportions; [statistical method as in outcome 1, analysis 1]

22. Secondary Outcome: Change From Baseline in Mini-Mental State Examination (MMSE) Total Scores at Week 12
Description: MMSE measured general cognitive functioning: orientation, memory, attention, calculation, language, visuospatial functions. Total score derived from sub-scores; total ranges from 0 - 30, higher score indicates better cognitive state. Change: mean score at Week 12 minus mean score at baseline.
Time Frame: baseline, Week 12
Population: Intent to Treat (ITT): (n=288; number of subjects responding)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Donepezil
Number analyzed (Participants) | 322
score on scale | 1.1 (2.75)
Statistical Analysis 1: Comparison: Donepezil; Change from baseline in total score at Week 12; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; One sample t-test, testing whether mean change from baseline is significantly different from zero

23. Secondary Outcome: Last Observation Carried Forward (LOCF) Change From Baseline in Mini-Mental State Examination (MMSE) Total Scores at Week 12
Description: as for outcome 22
Time Frame: baseline, Week 12 LOCF
Population: Intent to Treat (ITT) LOCF: (n=318; number of subjects responding)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Donepezil
Number analyzed (Participants) | 322
score on scale | 1.1 (2.79)
Statistical Analysis 1: Comparison: Donepezil; Change from baseline in total score at Week 12 Last Observation Carried Forward; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; One sample t-test, testing whether mean change from baseline is significantly different from zero

24. Secondary Outcome: Correlation Between Change From Baseline in Mini-Mental State Examination (MMSE) Score and Change From Baseline in Combined Patient and Caregiver Health Related Quality of Life (Alzheimer's Disease) (HR QoL-AD) Questionnaire Total Score
Description: MMSE cognitive function: Total 0 - 30, higher score, better cognitive state. Hr QoL- AD: physical health, energy, mood, living situation, memory, family, marriage, friends, chores, fun, money, self, and life as a whole using scale: 1 (poor) - 4 (excellent), possible total 13 - 52. Separate ratings from both patient and caregiver.
Time Frame: baseline, 12 Weeks
Population: Intent to Treat (ITT); n=207 (number of subjects who responded)
Measure: Number; unit: Pearson Product Correlation Coefficient
Arm/Group | Donepezil
Number analyzed (Participants) | 322
Pearson Product Correlation Coefficient | 0.33
Statistical Analysis 1: Comparison: Donepezil; Test type: Superiority or Other; p < 0.0001, correlation coefficient; P value tests whether Pearson Product Correlation Coefficient is significantly different from zero

25. Secondary Outcome: Correlation Between LOCF Change From Baseline in Mini-Mental State Examination (MMSE) Score and LOCF Change From Baseline in Combined Patient and Caregiver Health Related Quality of Life (Alzheimer's Disease) (HR QoL-AD) Questionnaire Total Score
Description: MMSE cognitive function. Total 0 - 30, higher score, better cognitive state. Hr QoL- AD: physical health, energy, mood, living situation, memory, family, marriage, friends, chores, fun, money, self, and life as a whole. Likert scale, 1 (poor) - 4 (excellent), possible total 13 to 52. Separate ratings from both the patient and the caregiver
Time Frame: baseline, Week 12 LOCF
Population: Intent to Treat (ITT) LOCF: (n=231; number of subjects responding).
Measure: Number; unit: Pearson Product Correlation Coefficient
Arm/Group | Donepezil
Number analyzed (Participants) | 322
Pearson Product Correlation Coefficient | 0.35
Statistical Analysis 1: Comparison: Donepezil; Test type: Superiority or Other; p < 0.0001, correlation coefficient; p-value tests whether Pearson Product Correlation Coefficient is significantly different from zero

26. Secondary Outcome: Change From Baseline in Combined Patient and Caregiver Health Related Quality of Life (Alzheimer's Disease) (HR QoL-AD) Questionnaire Total Scores
Description: Hr QoL- AD: physical health, energy, mood, living situation, memory, family, marriage, friends, chores, fun, money, self, and life as a whole. Likert scale, 1 (poor) - 4 (excellent), possible total 13 to 52. Separate ratings from both the patient and the caregiver. Change: mean score at Week 12 minus mean score at baseline.
Time Frame: baseline, 12 Weeks
Population: Intent to Treat (ITT). (n= 207; number of subjects who responded)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Donepezil
Number analyzed (Participants) | 322
score on scale | 1.4 (3.36)
Statistical Analysis 1: Comparison: Donepezil; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; One sample t-test, testing whether mean change from baseline is significantly different from zero

27. Secondary Outcome: LOCF Change From Baseline in Combined Patient and Caregiver Health Related Quality of Life (Alzheimer's Disease) (HR QoL-AD) Questionnaire Total Scores
Description: as for outcome 26
Time Frame: baseline, 12 Week LOCF
Population: Intent to Treat (ITT)LOCF: (n=231; number of subjects responding)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Donepezil
Number analyzed (Participants) | 322
score on scale | 1.4 (3.44)
Statistical Analysis 1: Comparison: Donepezil; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; One sample t-test, testing whether mean change from baseline is significantly different from zero

28. Secondary Outcome: Correlation Analysis: Change From Baseline in Combined Patient and Caregiver Quality of Life in Alzheimer's Disease(QoL-AD) Questionnaire Total Score Versus Number of Treatment Emergent Adverse Events (TEAEs)
Description: QoL- AD: physical health, energy, mood, living situation, memory, family, marriage, friends, chores, fun, money, self, and life as a whole. Likert scale, 1 (poor) - 4 (excellent), possible total 13 to 52. Patient and the caregiver totals combined and correlated to number of treatment emergent adverse events.
Time Frame: baseline, 12 Weeks
Population: Intent to Treat (ITT). (n=207 number of subjects responding)
Measure: Number; unit: Pearson Product Correlation Coefficient
Arm/Group | Donepezil
Number analyzed (Participants) | 322
Pearson Product Correlation Coefficient | -0.13
Statistical Analysis 1: Comparison: Donepezil; Test type: Superiority or Other; p = 0.0713, correlation coefficient

29. Secondary Outcome: Correlation Analysis: LOCF Change From Baseline in Combined Patient and Caregiver Quality of Life in Alzheimer's Disease (QoL-AD) Questionnaire Total Score Versus the Number of Treatment Emergent Adverse Events (TEAEs)
Description: QoL- AD: physical health, energy, mood, living situation, memory, family, marriage, friends, chores, fun, money, self, and life as a whole. Likert scale, 1 (poor) - 4 (excellent), possible total 13 to 52. Ratings from patient and the caregiver combined and correlated with number of treatment emergent adverse events.
Time Frame: baseline, 12 Weeks LOCF
Population: Intent to Treat (ITT) LOCF: (n=231; number of patients responding)
Measure: Number; unit: Pearson Product Correlation Coefficient
Arm/Group | Donepezil
Number analyzed (Participants) | 322
Pearson Product Correlation Coefficient | -0.15
Statistical Analysis 1: Comparison: Donepezil; Test type: Superiority or Other; p = 0.0225, Correlation coefficient

30. Secondary Outcome: Change From Baseline Total Score in EuroQuality of Life-5 Domains (EQoL-5D)
Description: EQoL-5D: measures index of health and defines it in 5 Domains:mobility,self-care,usual activities, pain/discomfort, anxiety/depression. Each domain evaluated on 3-point scale yielding 243 potential combinations; converted to utility values ranging from -0.59(worst state) to 1 (perfect state). Change: Week 12 mean score minus baseline mean score
Time Frame: baseline, 12 Weeks
Population: Intent to Treat (ITT) (n=290; number of subjects responding)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Donepezil
Number analyzed (Participants) | 322
score on scale | 0.015 (0.1071)
Statistical Analysis 1: Comparison: Donepezil; Test type: Superiority or Other; p = 0.0152, t-test, 2 sided; One sample t-test, testing whether mean change from baseline is significantly different from zero

31. Secondary Outcome: LOCF Change From Baseline Total Score in EuroQuality of Life-5 Domains (EQoL-5D)
Description: EQoL-5D: measures index of health & defines it in 5 Domains: mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each evaluated on 3-point scale yielding 243 potential combinations converted to utility values ranging from -0.59(worst state) to 1 (perfect state). Change:Week 12 mean score minus baseline mean score
Time Frame: baseline, 12 Weeks LOCF
Population: Intent to Treat (ITT) LOCF: (n=321; number of subjects responding)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Donepezil
Number analyzed (Participants) | 322
score on scale | 0.013 (0.1053)
Statistical Analysis 1: Comparison: Donepezil; Test type: Superiority or Other; p = 0.0229, t-test, 2 sided; One sample t-test, testing whether mean change from baseline is significantly different from zero

32. Secondary Outcome: Change From Baseline in Visual Analog Scale (VAS) of Subject's Overall Health Included in EuroQuality of Life-5 Domains (EQoL-5D)Questionnaire
Description: EuroQuality of Life-5 Domains (EQoL-5D)Questionnaire includes a visual analogue scale (VAS) of subject's overall health with 0 (worst state) to 100 (best state). Change: mean score at Week 12 minus mean score at baseline.
Time Frame: baseline, 12 Weeks
Population: Intent to Treat (ITT): (n=286; number of subjects responding).
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Donepezil
Number analyzed (Participants) | 322
score on scale | 3.7 (10.55)
Statistical Analysis 1: Comparison: Donepezil; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; One sample t-test, testing whether mean change from baseline is significantly different from zero

33. Secondary Outcome: LOCF Change From Baseline in Visual Analog Scale (VAS) of Subject's Overall Health Included in EuroQuality of Life-5 Domains (EQoL-5D) Questionnaire
Description: EuroQuality of Life-5 Domains (EQoL-5D) Questionnaire includes a visual analogue scale (VAS) of subject's overall health with 0 (worst state) to 100 (best state). Change: mean score at Week 12 minus mean score at baseline.
Time Frame: baseline, 12 Weeks LOCF
Population: Intent to Treat (ITT)LOCF: (n=318; number of subjects responding).
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Donepezil
Number analyzed (Participants) | 322
score on scale | 3.1 (10.91)
Statistical Analysis 1: Comparison: Donepezil; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; One sample t-test, testing whether mean change from baseline is significantly different from zero

34. Secondary Outcome: Change From Baseline in Subject's Mobility at Week 12
Description: EuroQuality of Life-5 Domains: health related tool (not disease specific) measuring index of health & defines health in 5 Domains, including mobility (no problem walking, some problems walking, confined to bed). Analysis of difference between the number of subjects with "any problem" and "no problem" at baseline versus at Week 12.
Time Frame: baseline, 12 Weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Donepezil
Number analyzed (Participants) | 322
participants
  Any Problem | 129
  No Problem | 161
Statistical Analysis 1: Comparison: Donepezil; Test type: Superiority or Other; p = 0.7963, McNemar; McNemar's Test for paired proportions tested the difference between the proportion of subjects with "Any problem" at baseline versus Week 12

35. Secondary Outcome: Change From Baseline in Subject's Mobility at Week 12 LOCF
Description: EuroQuality of Life-5 Domains: health related tool (not disease specific) measuring index of health & defines health in 5 Domains, including mobility (no problem walking, some problems walking, confined to bed). Analysis of difference between the proportion of subjects with "any problem" at baseline versus Week 12 LOCF
Time Frame: Week 12 LOCF
Population: Intent to Treat (ITT) LOCF: All Subjects who did not have a response for post baseline assessment were not included in analysis
Measure: Number; unit: Participants
Arm/Group | Donepezil
Number analyzed (Participants) | 322
Participants
  Any Problem | 147
  No Problem | 174
Statistical Analysis 1: Comparison: Donepezil; Test type: Superiority or Other; p = 1.0000, McNemar; McNemar's Test for paired proportions tested the difference between the proportion of subjects with "Any problem" at baseline versus Week 12 LOCF

36. Secondary Outcome: Change From Baseline in Subject's Self-Care at Week 12
Description: EuroQuality of Life-5 Domains: health related tool (not disease specific) measuring index of health & defines health in 5 Domains, including self-care (no problem, some problems, unable to wash or dress). Analysis of difference between the number of subjects with "any problem" and "no problem" at baseline versus at Week 12
Time Frame: baseline, Week 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Donepezil
Number analyzed (Participants) | 322
participants
  Any Problem | 122
  No Problem | 168
Statistical Analysis 1: Comparison: Donepezil; Test type: Superiority or Other; p = 0.0719, McNemar; [statistical method as in outcome 34, analysis 1]

37. Secondary Outcome: Change From Baseline in Subject's Self-Care at Week 12 LOCF
Description: EuroQuality of Life-5 Domains: health related tool (not disease specific) measuring index of health & defines health in 5 Domains, including self-care (no problem, some problems, unable to wash or dress). Analysis of difference between the number of subjects with "any problem" and "no problem" at baseline versus at Week 12 LOCF.
Time Frame: baseline, 12 Weeks LOCF
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Donepezil
Number analyzed (Participants) | 322
Participants
  Any Problem | 140
  No Problem | 181
Statistical Analysis 1: Comparison: Donepezil; Test type: Superiority or Other; p = 0.1779, McNemar; [statistical method as in outcome 35, analysis 1]

38. Secondary Outcome: Change From Baseline in Subject's Usual Activities at Week 12
Description: EuroQuality of Life-5 Domains: health related tool (not disease specific) measuring index of health & defines health in 5 Domains, including usual activities(no problem, some problem, unable to perform). Analysis of difference between the number of subjects with "any problem" and "no problem" at baseline versus at Week 12.
Time Frame: baseline, Week 12
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Donepezil
Number analyzed (Participants) | 322
Participants
  Any Problem | 181
  No Problem | 109
Statistical Analysis 1: Comparison: Donepezil; Test type: Superiority or Other; p = 1.0000, McNemar; [statistical method as in outcome 34, analysis 1]

39. Secondary Outcome: Change From Baseline in Subject's Usual Activities at Week 12 LOCF
Description: EuroQuality of Life-5 Domains: health related tool (not disease specific) measuring index of health & defines health in 5 Domains, including usual activities (no problem, some problem, unable to perform). Analysis of difference between the number of subjects with "any problem" and "no problem" at baseline versus at Week 12 LOCF
Time Frame: baseline, 12 Weeks LOCF
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Donepezil
Number analyzed (Participants) | 322
Participants
  Any Problem | 203
  No Problem | 118
Statistical Analysis 1: Comparison: Donepezil; Test type: Superiority or Other; p = 0.8575, McNemar; [statistical method as in outcome 35, analysis 1]

40. Secondary Outcome: Change From Baseline in Subject's Pain/Discomfort at Week 12
Description: EuroQuality of Life-5 Domains: health related tool (not disease specific) measuring index of health & defines health in 5 Domains, including discomfort(no pain, moderate pain, extreme pain). Analysis of difference between the number of subjects with "any problem" and "no problem" at baseline versus at Week 12.
Time Frame: baseline, Week 12
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Donepezil
Number analyzed (Participants) | 322
Participants
  Any Problem | 147
  No Problem | 143
Statistical Analysis 1: Comparison: Donepezil; Test type: Superiority or Other; p = 1.0000, McNemar; [statistical method as in outcome 34, analysis 1]

41. Secondary Outcome: Change From Baseline in Subject's Pain/Discomfort at Week 12 LOCF
Description: EuroQuality of Life-5 Domains: health related tool (not disease specific) measuring index of health & defines health in 5 Domains, including discomfort(no pain, moderate pain, extreme pain). Analysis of difference between the proportion of subjects with "any problem" at baseline versus Week 12 LOCF
Time Frame: Week 12 LOCF
Population: Intent to Treat (ITT)LOCF: All Subjects who did not have a response for post baseline assessment were not included in analysis
Measure: Number; unit: Participants
Arm/Group | Donepezil
Number analyzed (Participants) | 322
Participants
  Any Problem | 162
  No Problem | 159
Statistical Analysis 1: Comparison: Donepezil; Test type: Superiority or Other; p = 1.0000, McNemar; [statistical method as in outcome 35, analysis 1]

42. Secondary Outcome: Change From Baseline in Subject's Anxiety/Depression at Week 12
Description: EuroQuality of Life-5 Domains: health related tool (not disease specific) measuring index of health & defines health in 5 Domains, including anxiety/depression(none, moderate or extreme anxiety/depression). Analysis of difference between the number of subjects with "any problem" and "no problem" at baseline versus at Week 12.
Time Frame: baseline, Week 12
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Donepezil
Number analyzed (Participants) | 322
Participants
  Any Problem | 158
  No Problem | 132
Statistical Analysis 1: Comparison: Donepezil; Test type: Superiority or Other; p = 0.0131, McNemar; [statistical method as in outcome 34, analysis 1]

43. Secondary Outcome: Change From Baseline in Subject's Anxiety/Depression at Week 12 LOCF
Description: EuroQuality of Life-5 Domains: health related tool (not disease specific) measuring index of health & defines health in 5 Domains, including anxiety/depression (none, moderate or extreme anxiety/depression). Analysis of difference between the proportion of subjects with "any problem" and "no problem" at baseline versus at Week 12 LOCF
Time Frame: baseline, Week 12 LOCF
Population: as for outcome 41
Measure: Number; unit: Participants
Arm/Group | Donepezil
Number analyzed (Participants) | 322
Participants
  Any Problem | 179
  No Problem | 142
Statistical Analysis 1: Comparison: Donepezil; Test type: Superiority or Other; p = 0.0078, McNemar; [statistical method as in outcome 35, analysis 1]

ADVERSE EVENTS:
Arm/Group | Donepezil
Serious Adverse Events (participants affected / at risk) | 12
Other Adverse Events (participants affected / at risk) | 54
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Donepezil
Death (General disorders) | 4/370
Bradycardia (Cardiac disorders) | 1/370
Diverticulum (Gastrointestinal disorders) | 1/370
Cholecystitis (Hepatobiliary disorders) | 1/370
Diverticulitis (Infections and infestations) | 1/370
Lobar Pneumonia (Infections and infestations) | 1/370
Pneumonia (Infections and infestations) | 1/370
Urinary Tract Infection (Infections and infestations) | 1/370
Urosepsis (Infections and infestations) | 1/370
Hypercalcaemia (Metabolism and nutrition disorders) | 1/370
Hypoglycemia (Metabolism and nutrition disorders) | 1/370
Lung Neoplasm Maglinant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/370
Cerebrovascular Accident (Nervous system disorders) | 1/370
Syncope (Nervous system disorders) | 1/370
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Donepezil
Diarrhoea (Gastrointestinal disorders) | 13/370
Nausea (Gastrointestinal disorders) | 22/370
Vomiting (Gastrointestinal disorders) | 12/370
Asthenia (General disorders) | 8/370
Headache (Nervous system disorders) | 13/370
Insomnia (Psychiatric disorders) | 9/370

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other